CLINICAL TRIAL: NCT02917148
Title: MicroRNAs as Diagnostic and Predictive Biomarkers for Acute Graft Versus Host Disease
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Funding
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Cheryl Mensah, MD, Northwell Health
Other Study IDs: 15-229
Record Dates: First submitted 2016-09-21; First posted 2016-09-28 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2016-09

CONDITIONS: Acute GVH Disease
MeSH Terms: interventions — Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This blood will be collected in lavender top, EDTA tubes; some plasma (or serum) may be collected and stored for additional analysis.
  Plasma and serum samples from all patients will be frozen at -20 o C immediately after collection. RNAs will be extracted from plasma using Ambion RecoverAll kits, according to the directions provided by the manufacturer. Quantitative reverse-transcriptase polymerase chain reaction (qRT-PCR) will be performed on the samples as well. 754 microRNAs will be tested using ABI OpenArray platform.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aGVHD: Patient who undergo allogeneic transplant with clinical and/or biopsy-proven diagnosis of aGVHD within the first 100 days post-transplant.
  Interventions: Other: Peripheral Venipuncture or Blood draw from Central Line
- non aGVHD: Patients who undergo allogeneic transplant but do not develop aGVHD.

INTERVENTIONS:
Other: Peripheral Venipuncture or Blood draw from Central Line
  Other Names: Venipuncture; Blood Draw
  Groups: aGVHD

SUMMARY:
The goal of this research proposal is to identify a miRNA expression profile as a biomarker to diagnose and predict acute graft versus host disease (aGVHD) in patients who undergo allogeneic transplantation. This biomarker, once identified, will need validation in larger cohorts.

DETAILED DESCRIPTION:
Human subjects that volunteer to participate in this study will be requested to have approximately 20 cc of blood drawn (about 12 tablespoons) at several time intervals. These time intervals include prior to conditioning regimen for transplant, the day of transplantation, day +30, +60 and +100 after transplantation. If a given subject develops acute graft-versus-host disease, a blood sample will be obtained at that time as well. The amount of blood samples collected in an 8 week period will not exceed 50 ml and collection will not occur more than twice a week. There will be no pregnant women or children involved in the investigators study.

All patients involved in the study will be undergoing bone marrow transplant and pregnancy screening is done in pre-transplant testing. This blood will be collected in lavender top, EDTA tubes; some plasma (or serum) may be collected and stored for additional analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fully matched allogeneic PBCSC and bone marrow transplantation who present with clinical signs and symptoms of grade II- IV aGVHD within 100 days after transplantation as defined by skin, GI, and/or liver involvement that are confirmed by biopsy, regardless of age
* Patients undergoing a matched, unrelated donor (8/8) or matched, related donor transplant (6/6)
* Allogeneic transplant is from donor's peripheral blood stem cells or bone marrow transplant
* Patients who develop grade II-IV aGVHD

Exclusion Criteria:

* Patients who receive transplants from incompletely matched donors
* Patients who receive T cell depleted transplants
* Patients who receive haplo-identical transplants
* Pregnant Patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients included in the study will be patients undergoing allogeneic transplantation, and some will suffer from aGVHD and some will not.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Identify plasma microRNA expression in stem cell transplant patients with acute graft versus host disease compared to controls. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Mensah, MD, Principal Investigator — Northwell Health
Locations (1):
- Monter Cancer Center, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferrara JL, Levine JE, Reddy P, Holler E. Graft-versus-host disease. Lancet. 2009 May 2;373(9674):1550-61. doi: 10.1016/S0140-6736(09)60237-3. Epub 2009 Mar 11. PMID 19282026
- [Result] Paczesny S. Discovery and validation of graft-versus-host disease biomarkers. Blood. 2013 Jan 24;121(4):585-94. doi: 10.1182/blood-2012-08-355990. Epub 2012 Nov 19. PMID 23165480
- [Result] Xiao B, Wang Y, Li W, Baker M, Guo J, Corbet K, Tsalik EL, Li QJ, Palmer SM, Woods CW, Li Z, Chao NJ, He YW. Plasma microRNA signature as a noninvasive biomarker for acute graft-versus-host disease. Blood. 2013 Nov 7;122(19):3365-75. doi: 10.1182/blood-2013-06-510586. Epub 2013 Sep 16. PMID 24041574
- [Result] Xie LN, Zhou F, Liu XM, Fang Y, Yu Z, Song NX, Kong FS. Serum microRNA155 is increased in patients with acute graft-versus-host disease. Clin Transplant. 2014 Mar;28(3):314-23. doi: 10.1111/ctr.12314. Epub 2014 Feb 4. PMID 24494749